CLINICAL TRIAL: NCT04560621
Title: Managed Problem Solving for ART Adherence and HIV Care Retention Delivered by Community Health Workers: A Stepped Wedge Hybrid Type II Effectiveness Implementation Trial
Brief Title: Managed Problem Solving for ART Adherence and HIV Care Retention Delivered by Community Health Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Florence Momplaisir, MD, Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 843553
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAPS+ (Experimental)
  Interventions: Behavioral: Managed Problem Solving (MAPS)
- Standard of Care (No Intervention)

INTERVENTIONS:
Behavioral: Managed Problem Solving (MAPS) — MAPS is an individual-level, problem-solving intervention delivered in person and via telephone calls to HIV clinic patients. The intervention focuses on improving medication adherence through an iterative, five-step process which consists of 1) identifying barriers to adherence, 2) brainstorming to generate potential solutions, 3) decision-making and developing a plan of action, 4) implementing the plan, and 5) evaluating and modifying the plan as necessary. In-person sessions include education related to the treatment regimen and to common medication misperceptions; problem-solving to identify daily routines, cues, cognitive aids and social supports; screening to identify barriers related to depression, substance use, toxicity management and competing demands; and review of adherence data to determine where problems have occurred and to develop solutions.
  Arms: MAPS+

SUMMARY:
The Managed Problem Solving (MAPS) behavioral intervention is an EBP for behavior change in people living with HIV (PLWH). The investigators propose that MAPS can be delivered by trained Community Health Workers (CHWs). The use of CHWs to deliver MAPS is justified by their ability to develop trusting relationships with their clients and the need for task shifting in busy clinics. In order to also address retention in care, the investigators will adapt MAPS to also focus on problem solving activities tailored toward retention in care (now termed MAPS+). CHWs will be located in clinics to implement MAPS+ to improve viral suppression and care retention in PLWH. Data-to-care allows for identification of people who are lost to care and link these patients back to care. Currently, medication adherence and retention in HIV care are not targeted in data-to-care so the investigators will build on this approach to facilitate the identification of PLWH who are out of care and not virally suppressed to offer them MAPS+. The set of implementation strategies include task-shifting the delivery of MAPS+ to CHWs, providing the CHWs training and ongoing support, and increasing communication between the CHWs and medical care team via standardized protocols. The investigators will conduct a hybrid type II effectiveness-implementation trial with a stepped-wedge cluster randomized design in 12 clinics to test MAPS+ compared to usual care using a set of implementation strategies that will best support implementation. Each clinic will be randomized to one of three implementation start times. Baseline (usual care) data will be collected from each clinic for 6 months, followed by MAPS+ and the package of implementation strategies for 12 months, in three cohorts of 4 clinics each. Aim 1 will test the effectiveness of MAPS+ on clinical effectiveness outcomes, including viral suppression (primary) and retention (secondary). Aim 2 will examine the effect of the package of implementation strategies on reach. Implementation cost will also be measured. Aim 3 will apply a qualitative approach to understand processes, mechanisms, and sustainment of the implementation approach. The results will guide future efforts to implement behavioral EBPs across the HIV care continuum, consistent with the "treat" pillar of EHE, and move the science of implementation services, consistent with NIH strategic priorities.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* a man or woman living with HIV
* not retained in care and/or virally suppressed in year prior to trial initiation

Exclusion Criteria:

- incarcerated during the duration of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Undetectable HIV viral load (<20 copies/ml) | One year
  It is defined as having a viral load <20 copies/mL using the last available viral load at the end of one year (+/-60 days ) since trial initiation. VLs will be abstracted from the electronic medical record along with the date of lab collection.

SECONDARY OUTCOMES:
Adherence to HIV therapy | One year
  It is defined as the percentage of prescribed doses taken over 4 months and is calculated by dividing the observed pill-taking events by the number of doses prescribed for the study period.
Retention in care | One year
  It consists of having ≥1 visit with an HIV provider in each 6-month interval of the follow-up year with ≥60 days between clinic visits.
CD4 Count | One year
  It is defined as the measure of CD4 cells using the last available measure since trial initiation.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Cooper Early Intervention Program and Infectious Diseases, Camden, New Jersey
  - The Drexel Partnership Comprehensive Care Practice, Philadelphia, Pennsylvania
  - MacGregor Infectious Diseases Clinic at the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center Infectious Diseases Specialty Clinic at the University of Pennsylvania, Philadelphia, Pennsylvania
  - Jefferson HIV Ambulatory Care Program, Philadelphia, Pennsylvania
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - PHMC Care Clinic, Philadelphia, Pennsylvania
  - Temple Comprehensive HIV Program, Philadelphia, Pennsylvania
  - Einstein Immunodeficiency Center, Philadelphia, Pennsylvania
  - Mazzoni Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Van Pelt AE, Bilker WB, Nkwihorez H, Ghadimi F, Brady KA, Cidav Z, Schriger SH, Beidas RS, Gross R, Momplaisir F. Increasing antiretroviral therapy adherence and retention in care among adults living with HIV in Philadelphia: a study protocol for a stepped-wedge cluster-randomised type 2 hybrid effectiveness-implementation trial of managed problem-solving plus (MAPS+) delivered by community health workers. BMJ Open. 2023 Oct 21;13(10):e079585. doi: 10.1136/bmjopen-2023-079585. PMID 37865411